CLINICAL TRIAL: NCT05609968
Title: An Open-label, Multicenter, Phase 3 Randomized, Active-Comparator-Controlled Clinical Study of Pembrolizumab (MK-3475) in Combination With Sacituzumab Govitecan Versus MK-3475 Monotherapy as First-line Treatment in Participants With PD L1 TPS Greater Than or Equal to 50% Metastatic Non-small Cell Lung Cancer (KEYNOTE D46/EVOKE-03)
Brief Title: Study of Pembrolizumab (MK-3475) Monotherapy Versus Sacituzumab Govitecan in Combination With Pembrolizumab for Participants With Metastatic Non-small Cell Lung Cancer (NSCLC) With Programmed Cell Death Ligand 1 (PD-L1) Tumor Proportion Score (TPS) ≥50% (MK-3475-D46)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-D46; MK-3475-D46 (Other: MSD); PHRR230203-005387 (Registry Identifier: Philippine Health Research Registry (PHRR)); jRCT2031230031 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-503501-11-00 (Registry Identifier: EU CT); U1111-1287-4239 (Registry Identifier: UTN); 2022-000836-49 (EudraCT Number)
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death-2 (PD2, PD-2); Programmed Death-Ligand 2 (PDL2, PD-L2); Trophoblast Cell Surface Antigen-2 (TROP-2); Antibody-Drug Conjugate (ADC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Sacituzumab Govitecan (Experimental): Participants receive sacituzumab govitecan 10mg/kg intravenous (IV) infusion once weekly on Day 1 and Day 8 of a continuous 21-day cycle until progressive disease (PD) requiring discontinuation, unacceptable toxicity, withdrawal of consent, or death. Participants receive pembrolizumab 200mg IV infusion on Day 1 every 3 weeks (Q3W) for up to 35 cycles (each cycle length = 21 days).
  Interventions: Biological: Sacituzumab Govitecan; Biological: Pembrolizumab
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200mg IV infusion on Day 1 Q3W for up to 35 cycles (each cycle length = 21 days).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Sacituzumab Govitecan — IV infusion
  Other Names: Trodelvy®
  Arms: Pembrolizumab + Sacituzumab Govitecan
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda®

SUMMARY:
The purpose of this study is to compare pembrolizumab (MK-3475) in combination with sacituzumab govitecan with pembrolizumab alone with respect to progression-free survival (PFS) and overall survival (OS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR) among adults with metastatic non-small cell lung cancer (NSCLC) with programmed cell death ligand 1 (PD-L1) tumor proportion score (TPS) ≥50%).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a histologically or cytologically confirmed diagnosis of metastatic non-small cell lung cancer (NSCLC)
* Has confirmation that epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase 1 (ALK-1), or ROS proto-oncogene 1 (ROS-1)-directed therapy is not indicated as primary therapy
* Has provided tumor tissue that demonstrates PD-L1 tumor proportion score (TPS) ≥50% of tumor cells as assessed by immunohistochemistry (IHC) at a central laboratory
* Has a life expectancy of at least 3 months

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years
* Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC
* Has previously received treatment with Topoisomerase 1 inhibitors or Trop-2 targeted therapy
* Has received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti anti- programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received prior radiotherapy within 2 weeks of start of study intervention or has radiation-related toxicities requiring corticosteroids
* Has received radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks before study intervention administration
* Has cardiac disease

  * Myocardial infarction or unstable angina pectoris within 6 months of enrollment
  * History of serious ventricular arrhythmia, high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications; history of QT interval prolongation
  * New York Heart Association (NYHA) Class III or greater congestive heart failure or left ventricular ejection fraction of <40%
* Has active chronic inflammatory bowel disease
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab or sacituzumab govitecan and/or any of their excipients
* Has active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has history of human immunodeficiency virus (HIV) infection
* History of hepatitis B or known active hepatitis C virus infection
* Has history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2028-08-23 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 38 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as per the Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 is modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. PFS as assessed by blinded independent central review (BICR) will be presented.
Overall Survival (OS) | Up to approximately 48 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response (OR) | Up to approximately 38 months
  OR is defined as the confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by BICR.
Duration of Response (DOR) | Up to approximately 48 months
  DOR is defined as the time from the first documented evidence of a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until Progressive Disease (PD) or death due to any cause, whichever occurs first, in participants demonstrating a CR or PR. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Change from Baseline in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) | Baseline and up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" will be scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better overall health status. Per protocol, the change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Change from Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Baseline and up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better level of physical functioning. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in Role Functioning (Items 6-7) Combined Score on the EORTC QLQ-C30 | Baseline and up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a better level of role functioning. Change from baseline in the role functioning (EORTC QLQ-C30 Items 6-7) combined score will be presented.
Change from Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30 | Baseline and up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicates a worse level of dyspnea. The change from baseline in dyspnea (EORTC QLQ-C30 Item 8) score will be presented.
Change from Baseline in Cough Score (Item 31) on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 (EORTC QLQ-LC13) | Baseline and up to approximately 48 months
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate more frequent coughing and a worse outcome. The change from baseline in cough (EORTC QLQ-LC13 Item 31) score will be presented.
Change from Baseline in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 | Baseline and up to approximately 48 months
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate worse level of chest pain. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score will be presented.
Time to Deterioration (TTD) in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the EORTC QLQ-C30 | Up to approximately 48 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") will be scored on a 7-point scale (1=Very Poor to 7=Excellent). Higher scores indicate a better overall outcome. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-C30 Items 29 and 30 will be presented.
TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better level of physical functioning. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-C30 Items 1-5 will be presented.
TTD in Role Functioning (Items 6-7) Combined Score on the EORTC QLQ-C30 | Up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a better level of role functioning. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-C30 Items 6-7 will be presented.
TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30 11 | Up to approximately 48 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicates a worse level of dyspnea. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-C30 Item 8 will be presented.
TTD in Cough Score (Item 31) on the EORTC QLQ-LC13 | Up to approximately 48 months
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate more frequent coughing and a worse outcome. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-LC13 Item 31 will be presented.
TTD in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 | Up to approximately 48 months
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate worse level of chest pain. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-LC13 Item 40 will be presented.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 48 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study intervention. Per protocol, the number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due To an AE | Up to approximately 48 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study intervention. Per protocol, the number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (180):
- United States (16):
  - Infirmary Cancer Care ( Site 0418), Mobile, Alabama
  - Profound Research LLC ( Site 0444), Oceanside, California
  - Clermont Oncology Center ( Site 0421), Clermont, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 0417), Miami, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0416), Orange City, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0407), Marietta, Georgia
  - Our Lady of the Lake RMC ( Site 0424), Baton Rouge, Louisiana
  - Henry Ford Hospital ( Site 0412), Detroit, Michigan
  - Profound Research LLC ( Site 0440), Farmington Hills, Michigan
  - Allina Health Cancer Institute - Abbott Northwestern Hospital ( Site 0425), Minneapolis, Minnesota
  - Basil Clinical ( Site 0441), Inwood, New York
  - White Plains Hospital-Center for Cancer Care ( Site 0403), White Plains, New York
  - Kaiser Permanente Northwest-Central Interstate--Oncology ( Site 0408), Portland, Oregon
  - Oregon Health & Science University ( Site 0427), Portland, Oregon
  - Houston Methodist Hospital ( Site 0419), Houston, Texas
  - Central Texas Veterans health care ( Site 0414), Temple, Texas
- Australia (3):
  - Orange Hospital-Clinical Trials Unit ( Site 0600), Orange, New South Wales
  - Cancer Research SA-St Andrews Hospital ( Site 0603), Adelaide, South Australia
  - Frankston Hospital-Oncology and Haematology ( Site 0601), Frankston, Victoria
- Brazil (6):
  - CRIO - CENTRO REGIONAL INTEGRADO DE ONCOLOGIA ( Site 0320), Fortaleza, Ceará
  - Hospital Tacchini ( Site 0322), Bento Gonçalves, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo ( Site 0321), Passo Fundo, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 0317), Santa Cruz do Sul, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 0318), Barretos, São Paulo
  - A. C. Camargo Cancer Center ( Site 0324), São Paulo
- Canada (5):
  - BC Cancer Abbotsford-Medical Oncology ( Site 0433), Abbotsford, British Columbia
  - Southlake Health- Oncology Clinical Trials ( Site 0435), Newmarket, Ontario
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre ( Site 0430), Greenfield Park, Quebec
  - St. Marys Hospital Center-Oncology ( Site 0434), Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux-oncology ( Site 0431), Trois-Rivières, Quebec
- Chile (2):
  - Oncovida ( Site 0334), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0332), Santiago, Region M. de Santiago
- China (35):
  - Second Affiliated hospital of Anhui Medical University ( Site 0126), Hefei, Anhui
  - Anhui Provincial Hospital ( Site 0136), Hefei, Anhui
  - Beijing Cancer hospital ( Site 0104), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 0106), Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University ( Site 0105), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital-Medical Oncology ( Site 0130), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0131), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 0132), Xiamen, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 0125), Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University ( Site 0113), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 0119), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0127), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 0116), Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0115), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0107), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 0124), Changsha, Hunan
  - The Second Xiangya Hospital of Central South University ( Site 0135), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School ( Site 0112), Nanjing, Jiangsu
  - Nantong Tumor Hospital-Medical Oncology ( Site 0122), Nantong, Jiangsu
  - The First Affliated Hospital of Suzhou University ( Site 0114), Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University ( Site 0134), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 0117), Changchun, Jilin
  - Jilin Province Tumor Hospital-clinical research ( Site 0118), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University-Oncology ( Site 0133), Xi'an, Shaanxi
  - Jinan Central Hospital-oncology department ( Site 0121), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 0120), Linyi, Shandong
  - Shanghai Chest Hospital ( Site 0101), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center-Oncology ( Site 0102), Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University ( Site 0103), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 0129), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 0128), Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University ( Site 0109), Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine ( Site 0110), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 0111), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0108), Hangzhou, Zhejiang
- Estonia (2):
  - North Estonia Medical Centre Foundation-Chemotherapy ( Site 0621), Tallinn, Harju
  - Tartu University Hospital-Radiotherapy and oncology ( Site 0620), Tartu, Tartu
- Germany (7):
  - Universitätsmedizin Mannheim ( Site 0654), Mannheim, Baden-Wurttemberg
  - Klinikum Kempten ( Site 0655), Kempten (Allgäu), Bavaria
  - Klinikum Würzburg Mitte ( Site 0651), Würzburg, Bavaria
  - Katholisches Klinikum Koblenz ( Site 0650), Koblenz, Rhineland-Palatinate
  - Krankenhaus Martha-Maria Halle-Dölau-Klinik für Innere Medizin II ( Site 0657), Halle, Saxony-Anhalt
  - Vivantes Hospital Spandau-Klinik für Innere Medizin, Hämatologie, Onkologie und Gastroenterologie- ( Site 0656), Berlin
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf-Lungenklinik Heckeshorn ( Site 0653), Berlin
- Greece (3):
  - Errikos Dunant Hospital Center-Fourth Department of Oncology and Clinical Trials Unit ( Site 0141), Athens, Attica
  - Sotiria Thoracic Diseases Hospital of Athens-3rd Dept of Internal Medicine, Oncology Unit ( Site 0140), Athens, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 0142), Thessaloniki
- Israel (5):
  - Shaare Zedek Medical Center-Oncology ( Site 0176), Jerusalem
  - Meir Medical Center-oncology ( Site 0171), KfarSaba
  - Rabin Medical Center-Oncology ( Site 0174), Petah Tikva
  - Sourasky Medical Center-Oncology ( Site 0175), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 0179), Ẕerifin
- Italy (7):
  - Azienda Ospedaliera S. Giovanni Addolorata-Oncologia Medica ( Site 0677), Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII ( Site 0674), Bergamo, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0673), Milan, Lombardy
  - Azienda Ospedaliera Dei Colli-U.O.C Pneumologia Oncologica DH PNL ONC ( Site 0671), Naples, Napoli
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 0675), Florence, Tuscany
  - Casa di Cura Dott. Pederzoli-LUNG-UNIT TORACIC ( Site 0670), Peschiera del Garda, Verona
  - Azienda Ospedaliero Universitaria di Parma-UO Oncologia Medica ( Site 0676), Parma
- Japan (20):
  - Aichi Cancer Center ( Site 0018), Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center ( Site 0008), Matsuyama, Ehime
  - Kurume University Hospital ( Site 0014), Kurume, Fukuoka
  - Takarazuka City Hospital ( Site 0015), Takarazuka, Hyōgo
  - Kanazawa University Hospital ( Site 0019), Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center ( Site 0016), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 0001), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 0012), Sendai, Miyagi
  - Niigata Cancer Center Hospital ( Site 0017), Niigata, Niigata
  - Kurashiki Central Hospital ( Site 0011), Kurashiki, Okayama-ken
  - Kansai Medical University Hospital ( Site 0005), Hirakata, Osaka
  - Kindai University Hospital ( Site 0013), Sakai, Osaka
  - Saitama Prefectural Cancer Center ( Site 0002), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 0004), Nagaizumi-cho,Sunto-gun, Shizuoka
  - Tokyo Metropolitan Komagome Hospital ( Site 0020), Bunkyo Ku, Tokyo
  - National Hospital Organization Kyushu Medical Center ( Site 0009), Fukuoka
  - Kyushu University Hospital ( Site 0010), Fukuoka
  - Okayama University Hospital ( Site 0007), Okayama
  - Nippon Medical School Hospital ( Site 0003), Tokyo
  - Wakayama Medical University Hospital ( Site 0006), Wakayama
- Latvia (4):
  - Daugavpils Regional Hospital-Oncology Department ( Site 0194), Daugavpils, Daugavpils Novads
  - Liepjas reionl slimnca ( Site 0191), Liepāja
  - Pauls Stradins Clinical Univeristy Hospital-Chemotherapy department ( Site 0192), Riga
  - RIGA EAST UNIVERSITY HOSPITAL ,Oncology Centre of Latvia-Out-patient and Day patient facility of Ch ( Site 0193), Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos-Pulmonology ( Site 0692), Kaunas, Kaunas County
  - Vilnius University Hospital Santaros Clinics Affiliate - National Cancer Center ( Site 0691), Vilnius
- Malaysia (3):
  - Hospital Raja Perempuan Zainab II-Medical Department ( Site 0035), Kota Bharu, Kelantan
  - Hospital Pulau Pinang-Oncology, radiotherapy and palliat ( Site 0034), George Town, Pulau Pinang
  - Beacon Hospital Sdn Bhd ( Site 0033), Petaling Jaya, Selangor
- Mexico (6):
  - COI Tijuana - Centro Oncológico Internacional ( Site 0350), Tijuana, Estado de Baja California
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Servicio de Oncología ( Site 0352), Monterrey, Nuevo León
  - Medical Care and Research SA de CV ( Site 0353), Mérida, Yucatán
  - Centro de Investigacion Medica Aguascalientes ( Site 0340), Aguascalientes
  - Oaxaca Site Management Organization ( Site 0346), Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca ( Site 0351), Oaxaca City
- Peru (8):
  - Clinica Vallesur - AUNA ( Site 0360), Arequipa, Ariqipa
  - Instituto Regional de Enfermedades Neoplasicas del Centro (IREN CENTRO) ( Site 0362), Concepción, Departamento de Junín
  - Centro de investigacion Clínica Trujillo ( Site 0358), Trujillo, La Libertad
  - Clínica San Antonio ( Site 0366), Trujillo, La Libertad
  - Detecta Clínica ( Site 0364), Surquillo, Lima region
  - Clínica Internacional - Sede San Borja ( Site 0356), Lima
  - Instituto Neuro Cardiovascular de las Americas ( Site 0365), Lima
  - Hospital Cayetano Heredia ( Site 0361), Lima
- Philippines (3):
  - Metro Davao Medical and Research Center ( Site 0047), Davao City, Davao Del Sur
  - ST. LUKE'S MEDICAL CENTER ( Site 0046), Quezon City, National Capital Region
  - Cebu Doctors University Hospital ( Site 0045), Cebu
- Poland (7):
  - Med-Polonia Sp. z o. o. ( Site 0204), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 0208), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 0201), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 0200), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 0203), Przemyśl, Podkarpackie Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o. ( Site 0202), Prabuty, Pomeranian Voivodeship
  - Szpital Rejonowy im. dr. J. Rostka w Raciborzu ( Site 0207), Racibórz, Silesian Voivodeship
- Romania (6):
  - Gral Medical SRL-Medical Oncology ( Site 0220), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 0217), Cluj-Napoca, Cluj
  - Amethyst Radiotherapy Center-Oncologie Medicala ( Site 0216), Florești, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 0215), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 0219), Timișoara, Timiș County
  - Institutul Oncologic-Oncologie Medicala ( Site 0218), Cluj-Napoca
- South Korea (5):
  - Chonnam National University Hwasun Hospital-Pulmonology ( Site 0061), Hwasun, Jeonranamdo
  - Pusan National University Yangsan Hospital ( Site 0060), Pusan, Kyongsangnam-do
  - Chungnam national university hospital-Department of Internal Medicine ( Site 0063), Daejeon, Taejon-Kwangyokshi
  - Asan Medical Center ( Site 0064), Seoul
  - Korea University Guro Hospital-Internal Medicine ( Site 0062), Seoul
- Taiwan (7):
  - Chung Shan Medical University Hospital ( Site 0078), Taichung, Taichung
  - National Taiwan University Cancer Center (NTUCC) ( Site 0079), Taipei City, Taipei
  - E-Da hospital ( Site 0075), Kaohsiung City
  - China Medical University Hospital-Internal Medicine ( Site 0083), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 0076), Tainan
  - National Taiwan University Hospital-Internal Medicine ( Site 0080), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0082), Taoyuan District
- Thailand (6):
  - Bangkok Metropolitan Administration Medical College and Vajira Hospital ( Site 0097), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 0090), Bangkok, Bangkok
  - Lampang Cancer Hospital ( Site 0098), Lampang, Changwat Lampang
  - Songklanagarind hospital ( Site 0091), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0092), Muang, Chiang Mai
  - Sunpasitthiprasong Hospital ( Site 0093), Ubon Ratchathani
- Turkey (Türkiye) (8):
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 0265), Ankara
  - Liv Hospital Ankara-Oncology ( Site 0274), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 0268), Ankara
  - Trakya University-Medical Oncology ( Site 0270), Edirne
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi ( Site 0267), Istanbul
  - VM Medical Park Pendik Hospital ( Site 0271), Istanbul
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 0266), Izmir
  - Mersin Sehir Eğitim ve Araştırma Hastanesi ( Site 0275), Mersin
- United Kingdom (4):
  - Leicester Royal Infirmary-HOPE Clinical Trials Unit ( Site 0300), Leicester, Leicestershire
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 0302), London, London, City of
  - University College London Hospital ( Site 0305), London, London, City of
  - The Clatterbridge Cancer Centre ( Site 0303), Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26242&tenant=MT_MSD_9011